CLINICAL TRIAL: NCT01831726
Title: Modular Phase II Study to Link Targeted Therapy to Patients With Pathway Activated Tumors: Module 2 - Dovitinib for Patients With Tumor Pathway Activations Inhibited by Dovitinib Including Tumors With Mutations or Translocations of FGFR, PDGFR, VEGF, cKIT, FLT3, CSFR1, Trk and RET
Brief Title: Dovitinib for Patients With Tumor Pathway Activations Inhibited by Dovitinib
Acronym: SIGNATURE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258AUS26
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Tumor Pathway Activations Inhibited by Dovitinib
Keywords: Solid tumor malignancy; hematologic malignancy; mutation; translocations; FGFR; PDGFR; VEGF; cKIT; FLT3; CSR1; Trk; RET; TKI258; dovitinib; signature; AML; acute myelogenous leukemia; GIST; gastrointestinal stromal tumor; Head and Neck cancer; Melanoma; NSCLC; non-small cell lung carcinoma; lung cancer; ovarian cancer; thyroid cancer; amplification
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Gastrointestinal Stromal Tumors; Head and Neck Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Ovarian Neoplasms; Thyroid Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TKI258 (Experimental): Dovitinib (TKI) will be dosed on a flat scale of 500 mg on a 5 days on/2 days off dosing schedule.
  Interventions: Drug: Dovitinib (TKI258)

INTERVENTIONS:
Drug: Dovitinib (TKI258) — Dovitinib (TKI) will be dosed on a flat scale of 500 mg on a 5 days on/2 days off dosing schedule.

SUMMARY:
The purpose of this signal seeking study was to determine whether treatment with dovitinib (TKI258) demonstrated sufficient efficacy in select pathway-activated solid tumors and/or hematologic malignancies to warrant further study.

DETAILED DESCRIPTION:
This was a phase II, open label study to determine the efficacy and safety of treatment with dovitinib (TKI258) in patients with a diagnosis of select solid tumors or hematological malignancies that have been pre-identified (prior to study consent) to have mutations, translocations or amplifications and whose disease has progressed on or after standard treatment.

Genomic profiling is becoming more accessible to patients and their physicians. As such, more patients have been identified with potentially-actionable mutations, translocations or amplifications but do not have access to targeted drug treatment. This is a signal-seeking study to match patients with tumor pathway activations inhibited by dovitinib to the RTK inhibitor dovitinib. Pre-identification of mutations, translocations, or amplifications will be performed locally at a CLIA certified laboratory prior to participation on the trial.

For the purpose of this study, genomic profiling is not considered part of screening. Informed consent must be signed before any screening activities take place. Once eligibility (screening criteria met) has been confirmed by Novartis, the patient will initiate therapy with dovitinib single-agent. The patient may not receive any additional anti-cancer therapy during treatment with dovitinib.

Patients received study treatment until disease progression (assessed by investigator per RECIST 1.1 or appropriate hematologic response criteria), unacceptable toxicity, death or discontinuation from study treatment for any other reason (e.g., withdrawal of consent, start of a new anti-neoplastic therapy or at the discretion of the investigator), otherwise known as End of Treatment. All patients who discontinue from study treatment due to disease progression must have their progression clearly documented.

Disease assessment (by RECIST 1.1 or appropriate hematological response criteria) will be performed every 8 weeks (±4 days) after first dose of study drug (Day 1 of every odd cycle), until disease progression or end of treatment, whichever occurs first. The frequency of disease assessment may be reduced to every 12 weeks for patients who have at least 4 post-baseline disease assessments and are clinically stable (except AML patients). Scans was assessed locally by the investigator. After discontinuation of treatment, patients, regardless of reason for treatment discontinuation, will be followed for safety for 30 days after the last dose.

All patients will be followed for survival status every 3 months for 2 years after the last patient has enrolled in the study,regardless of treatment discontinuation reason (except if consent is withdrawn or patient is lost to follow-up)

ELIGIBILITY:
Key Inclusion Criteria:

Patients eligible for inclusion in this study had to meet all of the following criteria:

1. Patient's age was ≥ 18 years of age at the time of signing informed consent.
2. Patient had a confirmed diagnosis of a selected solid tumor (except for primary diagnosis of urothelial tumors, hepatocellular carcinoma (HCC), endometrial carcinoma, metastatic breast cancer (mBC), squamous NSCLC, and renal cell carcinoma (RCC)) or hematologic malignancies (except for primary diagnosis of FLT3 AML and multiple myeloma). Additional tumor types could be excluded during the course of the study in the case of early futility or success based upon an interim analysis or at the discretion of Novartis.
3. Patient was in need of treatment because of progression or relapse defined as:

   * radiological progression for solid tumor and lymphoma
   * for hematologic malignancies, measureable progression or relapse by appropriate criteria
4. Patients had pre-identified tumor with a mutation and/or translocation of one of the known kinase targets of dovitinib. The qualifying alteration were assessed and reported by a CLIA-certified laboratory. The mutations included:

   1. FGFR 1-3 (amplifications were also allowed)
   2. PDGFRα or PDGFRβ
   3. VEGFR1-2 (KDR)
   4. FLT3, cKIT (amplifications are also allowed),
   5. RET, TrkA (NTRK1), or CSF-1R
5. Patient had archival tissue available for submission to allow for molecular testing related to pathway activation. If the tissue was not available or not of sufficient quantity the patient was willing to undergo a fresh tumor biopsy to allow for this analysis. The sample was submitted prior to first study dose unless agreed upon between Novartis and the investigator.
6. Patient received at least one prior treatment for recurrent, metastatic and /or locally advanced disease and for whom no standard therapy options were anticipated to result in a durable remission.
7. Diffuse large B cell lymphoma only: Patient received or was ineligible for autologous or allogeneic stem cell transplant. This did not apply to patients with Mantle cell lymphoma or follicular lymphoma
8. Patients with measurable disease as per appropriate guidelines:

   a. Solid Tumors: by RECIST 1.1
9. Lymphoma: Patient had at least one measurable nodal lesion (≥2 cm) according to Cheson criteria (Cheson 2007). In case where the patient had no measurable nodal lesions ≥ 2 cm in the long axis at screening, then the patient had at least one measurable extra-nodal lesion.
10. Leukemia only: Relapsed/refractory leukemia for which no standard therapy options were anticipated to result in a durable remission:

    1. Acute myelogenous leukemia (AML) by World Health Organization (WHO) classification (except FLT3) or acute lymphoblastic leukemia (ALL) relapsed or refractory to standard chemotherapy; unsuitable for standard chemotherapy or unwilling to undergo standard chemotherapy. Philadelphia chromosome (Ph) positive ALL eligible if failed prior tyrosine-kinase inhibitor therapy.
    2. Age > 60 years with AML (except FLT3) not candidates for or have refused standard chemotherapy, excluding patients with acute promyelocytic leukemia (APL) or with favorable cytogenetic abnormalities.
    3. For patients with Chronic Myeloid Leukemia (CML) only accelerated and blast phase CML were allowed.
11. Patient with an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
12. Patient with a life expectancy of at least 16 weeks
13. All Patients were having adequate bone marrow as described below:

    1. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L (not applicable for leukemia patients).
    2. Platelets (PLT) ≥ 75 x 109/L (no platelet transfusion within past 14 days) (not applicable for leukemia patients).
    3. Hemoglobin (Hgb) ≥ 9 g/dl (not applicable for leukemia patients).
    4. International Normalized Ratio (INR) ≤ 1.5.
    5. Serum amylase and lipase ≤ upper limit of normal (ULN).
14. All patients had adequate organ function defined as described below:

    1. Potassium, calcium (corrected for serum albumin) and magnesium within normal limits (WNL). Supplementation was allowed to meet eligibility requirements. Bisphosphonates to treat malignant hypercalcemia WERE NOT allowed.
    2. Serum creatinine ≤ 1.5 x ULN or Serum creatinine >1.5 - 3 x ULN if

       * creatinine clearance by 24-hr urine was ≥ 30 mL/min/1.73m2 (≥50 mL/min/1.73m2 in the presence of proteinuria as defined by inclusion criterion #16 or
       * calculated creatinine clearance (CrCl) was ≥ 30 mL/min using the Cockroft- Gault equation CrCl = (140 - age in years) x (weight in kg) / (72 x serum creatinine in mg/dL) (if female, multiply the number by 0.85)
    3. Alanine aminotransferase (AST) and/or aspartate aminotransferase (ALT) ≤ 3.0 x upper limit of normal range (ULN)
    4. Total serum bilirubin within normal range (or ≤ 1.5 x ULN)
15. Urine dipstick reading: Negative for proteinuria or, if documentation of +1 results for protein on dipstick reading, then total urinary protein ≤ 500 mg and measured creatinine clearance ≥ 50 mL/min/1.73m2 from a 24 hour urine collection.
16. For Leukemia patients, peripheral blast counts < 50,000 blasts/mm3

Key Exclusion Criteria:

Patients eligible for this study did not meet any of the following criteria:

1. Patients who received prior treatment with dovitinib (TKI258).
2. Patients with a known hypersensitivity to dovitinib (TKI258) or to its excipients.
3. Patients with brain metastasis or history of brain metastasis or leptomeningeal carcinomatosis.
4. Patients with diarrhea ≥ CTCAE grade 2.
5. Patients with neuropathy ≥ CTCAE grade 2.
6. Patients with acute or chronic pancreatitis.
7. Patients with external biliary drains.
8. Patients with a history of pulmonary embolism (PE), or untreated deep venous thrombosis (DVT) ≤ 6 months prior to starting study drug. Note: Patients with recent DVT who were treated with therapeutic anti-coagulant agents for at least 6 weeks are eligible.
9. Patients with impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   1. History or presence of serious uncontrolled ventricular arrhythmias.
   2. Clinically significant resting bradycardia.
   3. LVEF assessed by either 2-D echocardiogram (ECHO) < 50% or lower limit of normal (whichever was the higher), or 2-D multiple gated acquisition scan (MUGA) < 45% or lower limit of normal (whichever was the higher).
   4. Any of the following within 6 months prior to starting study drug: myocardial infarction (MI), severe/unstable angina, coronary artery bypass graft (CABG), congestive heart failure (CHF), cerebrovascular accident (CVA), transient ischemic Attack (TIA).
   5. Uncontrolled hypertension defined by a SBP ≥ 160 mm Hg and/or DBP ≥ 100 mm Hg, with or without anti-hypertensive medication(s). Initiation or adjustment of antihypertensive medication(s) was allowed prior to study entry.
10. Patients with uncontrolled diabetes mellitus.
11. Patients with clinical evidence of active CNS leukemia.
12. Patient who received Allogeneic stem cell transplant and/or had active has graft-versus host disease (GVHD).
13. Patient received Autologous stem cell transplant within last 4 weeks.
14. Impairment of GI function or GI disease that could significantly alter the absorption of dovitinib (e.g. severe ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
15. Any other condition that was, in the Investigator's judgment, contraindicate patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g. infection/inflammation, intestinal obstruction, unable to swallow oral medication, social/psychological complications.
16. Patients who were treated with any hematopoietic colony-stimulating growth factors (e.g.,G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, could be continued. Restriction was not applicable for patients with Leukemia.
17. Patient who received chemotherapy or other anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, monoclonal antibodies or mitomycin-C) prior to starting study drug or who had not recovered to a grade 1 from side effects of such therapy (except for alopecia and neuropathy). Patients with leukemia could receive therapy with hydroxyurea and/or steroids for the purpose of cytoreduction but must discontinue use prior to first dose of study drug.
18. Patients who received the last administration of an anticancer small molecule therapy (e.g. sunitinib, sorafenib, pazopanib, axitinib, everolimus, temsirolimus, ridaforolimus) ≤ 2 weeks prior to starting study drug, or who had not recovered from the side effects of such therapy.
19. Patients not able to discontinue their current anti-cancer therapy prior to first dose of study drug.
20. Patients who received radiotherapy ≤ 4 weeks prior to starting the study drug or who had not recovered from radiotherapy-related toxicities (note: palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting study drug is allowed).
21. Patients who had undergone major surgery (e.g., intra-thoracic, intra-abdominal, intrapelvic) ≤ 4 weeks prior to starting study treatment or who had not recovered from side effects of such surgery.
22. Patient was currently receiving antiplatelet therapy of prasugrel or clopidogrel, or full dose anticoagulation treatment with therapeutic doses of warfarin. However, treatment with low doses of warfarin (e.g., ≤ 2 mg/day) or locally accepted low doses of acetylsalicylic acid (up to 100 mg daily) to prevent cardiovascular events or strokes was allowed.
23. Patients with another primary malignancy within 3 years prior to starting study treatment, with the exception of adequately treated basal cell carcinoma, squamous cell carcinoma or other non-melanomatous skin cancer, or in-situ carcinoma of the uterine cervix.
24. Cirrhosis of the liver or known hepatitis B or C infection that was either acute or was considered chronic because the virus did not become undetectable:

    1. Hepatitis C Virus (HCV) infection: acute or chronic infection as depicted by a positive HCV RNA testing (note: in a patient with known anti-HCV but with a negative test for HCV RNA, re-testing for HCV RNA 4-6 months later was requested to confirm the resolution of HCV infection).
    2. Hepatitis B Virus (HBV) infection: acute infection (HBsAg+ with or without HBeAg+ or detectable serum HBV DNA), HBV carriers as evidence by ongoing presence of HBsAg and detectable serum HBV DNA levels.
25. Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing was not mandatory).
26. Patients who received investigational agents within ≤ 5t1/2 of the agent (or ≤ 4 weeks when half-life was unknown) prior to starting study drug.
27. Patient with history of non-compliance to medical regimen.
28. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
29. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they were using highly effective methods of contraception (defined below). Highly effective contraception had to be used by both sexes (female patients and their male partners) during study treatment and for 30 days after the last doseof study medication.

    Highly effective contraception methods included:
    * Total abstinence (when this was in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post- ovulation methods) and withdrawal were not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment.

    In case of oophorectomy alone, only when the reproductive status of the woman was confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female patients on the study the vasectomized male partner was the sole partner for that subject.
    * Combination of the following (a+b):

      1. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
      2. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
30. Oral, implantable, or injectable hormone contraceptives might be affected by cytochrome P450 interactions, and were therefore not considered effective for this study Women of child-bearing potential (sexually mature women) who had not undergone a hysterectomy or who were not naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), were required to have a negative serum pregnancy test ≤ 14 days prior to starting study drug.
31. Post-menopausal women were allowed to participate in this study. Women were considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks prior to entry in the study. In the case of oophorectomy alone, only when the reproductive status of the woman was confirmed by follow up hormone level assessment, then she was considered not of child bearing potential.
32. Fertile males not willing to use contraception. Fertile males must use condom with spermicide. Highly effective contraception, as defined above, was to be used by both sexes (male patients and their female partners) during study treatment and for 90 days after the last dose of study medication and was not to father a child in this period. A condom was required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (49):
- United States (49):
  - Alabama Oncology, Birmingham, Alabama
  - Highlands Oncology Group SC, Fayetteville, Arkansas
  - PCR Oncology, Pismo Beach, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Rocky Mountain Cancer Centers Rocky Mountain Cancer Centers, Greenwood Village, Colorado
  - Whittingham Cancer Center Norwalk Hospital, Norwalk, Connecticut
  - Memorial Cancer Institute Memorial Healthcare System, Hollywod, Florida
  - Cancer Specialists of North Florida Cancer Specialists (2), Jacksonville, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Space Coast Medical Associates Space Coast Cancer Center, Titusville, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - NorthWest Georgia Oncology Centers NW Georgia Oncology, Marietta, Georgia
  - Lurie Children's Hospital of Chicago Developmental Therapeutics, Chicago, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Indiana University Indiana Univ. - Purdue Univ., Indianapolis, Indiana
  - Horizon Oncology Center Horizon Oncology Ctr., Lafayette, Indiana
  - St. Agnes Hospital St. Agnes Hospital (2), Baltimore, Maryland
  - University of Michigan Int. Medicine Oncology, Ann Arbor, Michigan
  - Minnesota Oncology Hematology, P.A. Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Billings Clinic Onc Dept, Billings, Montana
  - Southeast Nebraska Oncology Cancer Center, Lincoln, Nebraska
  - Comprehensive Cancer Centers of Nevada CCC of Nevada- Southwest (2), Las Vegas, Nevada
  - Waverly Hematology Oncology, Cary, North Carolina
  - Oncology Hematology Care, Inc. Oncology Hematology Care (2), Cincinnati, Ohio
  - Cleveland Clinic Foundation Cleveland Clinic (19), Cleveland, Ohio
  - St. Charles Cancer Center, Bend, Oregon
  - Oregon Health & Science University OHSU Knight Cancer Institute, Portland, Oregon
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Rhode Island Hosp. (2), Providence, Rhode Island
  - Gibbs Cancer Center & Research Institute Spartanburg Reg. Healthcare, Spartanburg, South Carolina
  - Chattanooga Oncology and Hematology Assoicates, PC Chattanooga Oncology, Chattanooga, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Sarah Cannon Research Institute Tennessee Oncology, Nashville, Tennessee
  - Austin Cancer Centers Austin Cancer Center (2), Austin, Texas
  - Texas Oncology Texas Oncology - Sammons, Dallas, Texas
  - Texas Oncology Midtown Texas Oncology, Dallas, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Oncology Consultants Oncology Group, Houston, Texas
  - MD Anderson Cancer Center/University of Texas MD Anderson Cancer Center (3), Houston, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Intermountain Medical Center Intermountain Healthcare, Murray, Utah
  - Virginia Cancer Specialists Virginia Cancer Specialists, Fairfax, Virginia
  - Providence Regional Cancer Partnership Providence Reg. Cancer (2), Everett, Washington
  - Evergreen Hematology & Oncology, Spokane, Washington
  - Northwest Medical Specialties Hematology/Oncology, Tacoma, Washington
  - Wenatchee Valley Medical Center Wenatchee Valley, Wenatchee, Washington
  - Yakima Valley Memorial Hospital North Star Lodge Cancer Center, Yakima, Washington
  - Aurora Research Institute, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Ctr.-Froedtert Hospital, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TKI258
Started | 80
Completed | 0
Not Completed | 80
Not completed — Adverse Event | 16
Not completed — Death | 7
Not completed — Disease Progression | 49
Not completed — Physician Decision | 1
Not completed — Subject/guardian decision | 7

BASELINE CHARACTERISTICS:
Arm/Group | TKI258
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR)
Description: CBR determined by investigator assessment for each tumor assessment & defined as responses of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) ≥ 16 wks. Confirmed CR/PR or SD prior to 16 wks,but discontinued prior to 16 wks for reasons other than progressive disease,will have their clinical benefit defined non-evaluable; confirmed CR/PR or SD prior to 16 wks,but progressed prior to 16 wks,will be considered not achieving clinical benefit;if CR/PR/SD occurred prior to 16 wks,but progressed at or after 16 wks without evidence of CR/PR/SD at or after 16 wks,will also be considered not achieving clinical benefit. CBR will be analyzed by comparing achieved CBR with a historical control rate of each tumor type,& if there is at least 90% probability that the response rate in a tumor type exceeds the historical rate,then the tumor type will be considered a success. CBR: CR+PR+SD the assessment criteria was RECIST 1.1
Time Frame: Week 16
Population: Full Analysis Set (FAS) included all patients who received at least one dose of study drug.
  FAS was used for the analysis of efficacy endpoints.
Measure: Number; unit: number of participants
Arm/Group | TKI258
Number analyzed (Participants) | 80
number of participants
  Complete response (CR) | 0
  Partial response (PR) | 1
  Stable disease (SD) | 10
  Clinical benefit rate (CBR) | 11

2. Secondary Outcome: Overall Response (OR) of Partial Response (PR) or Greater
Description: Overall Response (OR) of Partial Response (PR) or greater based on local investigator assessment. For patients with solid tumors, the assessment criteria will be RECIST 1.1 and will include responses of CR and/or PR. For hematologic tumors other appropriate hematological response criteria will apply and are included in the appendices. ORR: CR+PR
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: number of participants
Arm/Group | TKI258
Number analyzed (Participants) | 80
number of participants
  Complete response (CR) | 0
  Partial response (PR) | 1
  Overall response rate (ORR) | 1

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression free survival (PFS) is defined as the time from the date of first dose to the date of first documented disease progression or relapse or death due to any cause.
Time Frame: 36 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TKI258
Number analyzed (Participants) | 80
months | 2.4 [1.8 to 3.7]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from the date of first dose to the date of death due to any cause. If a patient is not known to have died, survival time will be censored at the date of the last contact
Time Frame: 36 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TKI258
Number analyzed (Participants) | 80
months | 13.5 [5.9 to 14.7]

ADVERSE EVENTS:
Arm/Group | TKI258
Serious Adverse Events (participants affected / at risk) | 32/80
Other Adverse Events (participants affected / at risk) | 78/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TKI258 (N=80)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Chest pain (General disorders) | 2
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 2
Bile duct obstruction (Hepatobiliary disorders) | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral thrombosis (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Angioedema (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TKI258 (N=80)
Anaemia (Blood and lymphatic system disorders) | 8
Lymphopenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Sinus tachycardia (Cardiac disorders) | 4
Lacrimation increased (Eye disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 12
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 26
Diarrhoea (Gastrointestinal disorders) | 51
Dry mouth (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 8
Dysphagia (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Haemorrhoids (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 47
Vomiting (Gastrointestinal disorders) | 35
Asthenia (General disorders) | 13
Fatigue (General disorders) | 56
Mucosal inflammation (General disorders) | 4
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 7
Pyrexia (General disorders) | 7
Pneumonia (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 7
Alanine aminotransferase increased (Investigations) | 16
Amylase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 19
Blood alkaline phosphatase increased (Investigations) | 23
Blood bilirubin increased (Investigations) | 7
Blood creatinine increased (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 17
Lipase increased (Investigations) | 8
Platelet count decreased (Investigations) | 4
Weight decreased (Investigations) | 18
White blood cell count decreased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 34
Dehydration (Metabolism and nutrition disorders) | 17
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 27
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 9
Hyponatraemia (Metabolism and nutrition disorders) | 12
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 9
Headache (Nervous system disorders) | 15
Neuropathy peripheral (Nervous system disorders) | 5
Anxiety (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 4
Proteinuria (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 5
Night sweats (Skin and subcutaneous tissue disorders) | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 14
Hypotension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.